CLINICAL TRIAL: NCT01575483
Title: Korean Post-marketing Surveillance for Onglyza®
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CV181-171
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with T2DM: Patients with diagnosis of type 2 diabetes mellitus (T2DM) initiating Onglyza® treatment within the approved indications will be enrolled
  Interventions: Drug: No Intervention (subjects were previously treated with Onglyza®)

INTERVENTIONS:
Drug: No Intervention (subjects were previously treated with Onglyza®) — No Intervention
  Other Names: saxagliptin

SUMMARY:
The purpose of this post-marketing surveillance is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and efficacy of Onglyza® so that the regulatory authority can manage the marketing approval properly.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who are at least 18 years of age
* Patients with diagnosis of T2DM initiating Onglyza® treatment within the approved indications in Korea

Exclusion Criteria:

* Indication which is not approved for Onglyza® in Korea
* Patients with contraindication for the use of Onglyza® (as clarified in Korean label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of type 2 diabetes mellitus initiating Onglyza® treatment within the approved indications will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 3433 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

PRIMARY OUTCOMES:
Adverse events occurrence | 30 days after last dose of study drug

SECONDARY OUTCOMES:
Number of Adverse Events and Serious Adverse Events | 30 days after last dose of study drug
Effectiveness of Onglyza® measured by Hemoglobin A1c (HbA1c), fasting plasma glucose (FPG) and 2-hr post-prandial glucose (2-hr PPG) comparing baseline data | Baseline (Week 0), 12 weeks and 24 weeks of registration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Research Site, Seoul, South Korea

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4125&filename=CSR_Synopsis_CV181_171.pdf